CLINICAL TRIAL: NCT04091230
Title: Prospective Patient Blinded Randomized Trial Comparing Biopsy Specimen Quality in a Novel Biopsy Needle and Actuator Compared to Todays Standard Tru Cut Needle and Actuator.
Brief Title: New Biopsy Needle - Evaluation of Prostate Biopsy Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018/283
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: biopsy quality
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: 20 patients eligible for prostate biopsy are randomized into 2 arms (10+10 patients) using either the novel needle and actuator device or standard tru cut needle and actuator device used in the clinic today. On average 12 biopsies are taken from each patient. Biopsy quality is evaluated by the pathologist blinded to device used.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and pathologist are unaware of which needle/device is used. TRUSbx are taken from behind the back of the patient enabling masking from the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- novel needle (Experimental): TRUSbx using the 18 gauge (G) 25 centimeter(cm) novel needle with 19 millimeter (mm) sample notch and a new actuator. 12 biopsies / patient.
  Interventions: Device: TRUSbx
- standard tru cut needle (Active Comparator): TRUSbx using a standard tru cut biopsy needle (Mermaid Medical M-biopsy 18G 25 cm biopsy needle with a 19 mm sample notch) in a standard actuator ( Moller Medical Blue RBG-1000-10-1000). 12 biopsies/ patient.
  Interventions: Device: TRUSbx

INTERVENTIONS:
Device: TRUSbx — Trans Rectal UltraSound guided Prostate Biopsy
  Other Names: prostate biopsy

SUMMARY:
Patient blinded randomized prospective trial evaluating prostate biopsy quality of a novel biopsy needle.

DETAILED DESCRIPTION:
Prostate biopsy is the golden standard for diagnose of prostate cancer. Transrectal prostate biopsy (TRUSbx) is the most widely used technique. Due to the transrectal path the biopsy needle will bring bacteria from the colon into tissue. The patent should always receive prophylactic antibiotics to reduce the risk of clinical infection. Infections related to transrectal prostate biopsy (TRUSbx) are increasing in parallel with rising antibiotic resistance.

The investigators have in an ex-vivo setting previously shown a drastic reduction in bacterial transfer across the colon wall using a novel biopsy needle designed to minimize bacterial transfer. Biopsy of prostatectomy specimen using the novel needle has shown biopsy quality equal to the tru cut biopsy needle used today.

This is the first human pilot aiming to evaluate if biopsy quality of the novel needle is equal to the reference tru cut biopsy needle in prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for prostate biopsy
* Signed informed written consent

Exclusion Criteria:

* None (other than general contra indications for prostate biopsy or patient not willing to participate)

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Biopsy
Enrollment: 20 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
prostate biopsy length (measured by pathologist) | within 21 days post biopsy
  Length of biopsy specimen in millimeters

SECONDARY OUTCOMES:
prostate biopsy fragmentation | within 21 days post biopsy
  The number of sections the biopsy specimen is made of
General appearance of biopsy assessed by pathologist (biopsy quality) | within 21 days post biopsy
  General quality of biopsy specimen on a scale from 0-3 (no biopsy, poor, good, excellent)
prostate biopsy length (measured in biopsy needle chamber) | within 21 days post biopsy
  Length of biopsy specimen in millimeters
prostate biopsy length (measured in after removal from biopsy chamber) | within 21 days post biopsy
  Length of biopsy specimen in millimeters

OTHER OUTCOMES:
patient experience / pain | at the time of rectal ultrasound probe insertion, estimated to a timeframe of 5-30 seconds.
  Numeric rating Pain Scale rating from 0-10
patient experience / pain | at the time of injection needle advancement and periprostatic injection of local anesthesia, estimated to a timeframe of 5-10 seconds
  Numeric rating Pain Scale rating from 0-10
patient experience / pain | at the time of biopsy sampling.
  Numeric rating Pain Scale rating from 0-10
14 day complications | 14 days
  Any complications related to the biopsy (example infection, bleeding)
30 day complications | 30 days
  Any complications related to the biopsy (example infection, bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Linder, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Helsingborg Hospital, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No